CLINICAL TRIAL: NCT04892602
Title: Fibromyalgia in Rheumatiod and Psoriatic Arthritis Patients:Relationshipwith Disease Activity and Serum Vitamin Dlevel
Brief Title: Fibromyalgia in Rheumatiod and Psoriatic Patients
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alshimaa Hamdey Khalaf, Alshimaa hamdy khalaf, Sohag University
Other Study IDs: Soh-Med-21-05-03
Record Dates: First submitted 2021-05-16; First posted 2021-05-19 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Fibromyalgia, Secondary
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rheumatiod arthritis patients
  Interventions: Diagnostic Test: Serum vitaminDlevel
- Psoaritic arthritis
  Interventions: Diagnostic Test: Serum vitaminDlevel
- Control group
  Interventions: Diagnostic Test: Serum vitaminDlevel

INTERVENTIONS:
Diagnostic Test: Serum vitaminDlevel — Investigate about fibromyalgia in psoiaritic and rheumatiod arthritis patients ...and assesment of seum vitamin D level

SUMMARY:
the study based on investigate for fibromyalgia among rheumatiod arthritis patient and psoriatic arthritis.....and to what extent gibromyalgia affect disease activity indices ....and its relation to serum Vitamin D level in those patients

ELIGIBILITY:
Inclusion Criteria:

- adult onset disease any patient diagnosed as rheumatiod arthritis and psoriatic arthritis above18years old

Exclusion Criteria:

* any other autoimmune diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Those patient who diagnosed as rheumatiod arthritis and psoriatic arthritis..assess serum vitamin D level
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Serum vitamin D level | One year
  Blood test to asses hypovitaminosis in these patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Serum Vitamin Dlevel Disease activity indice